CLINICAL TRIAL: NCT00435396
Title: A Phase I, Open-label, Vaccination Study to Evaluate the Safety and Immunogenicity of the GSK Biologicals Recombinant CMV gB Sub-unit Vaccine GSK1492903A in CMV-seronegative Healthy Male Adult Subjects
Brief Title: Study to Evaluate Safety and Immunogenicity of the GSK Bio CMV Vaccine in CMV-seronegative Healthy Male Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 108890; 109211 (Other: GSK)
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infections, Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: GSK Biologicals' Recombinant CMV gB Vaccine GSK1492903A

INTERVENTIONS:
Biological: GSK Biologicals' Recombinant CMV gB Vaccine GSK1492903A — Intramuscular injection, 3 doses

SUMMARY:
This will be the first time in humans (FTIH) study with the GSK Bio recombinant gB antigen to evaluate safety and immunogenicity of this CMV candidate vaccine with a proprietary GSK adjuvant system. The vaccine will be administered to young male healthy subjects at 0, 1 and 6 months. The trial will assess the safety and immunogenicity of the candidate CMV vaccine. An additional secondary objective of this trial is to identify and validate a test which will be able to differentiate between previous CMV infection and CMV vaccination. Subjects will be followed for a total of 2 years.

DETAILED DESCRIPTION:
The protocol posting has been amended to reflect changes as a consequence of an amendment to the protocol. The section impacted by the change is Key inclusion & exclusion criteria. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Male between, and including, 18 and 40 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* The subject consents to being informed of his CMV and HSV serostatus.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Seronegative for CMV.
* Previously completed routine childhood vaccinations to the best of his knowledge.

Exclusion Criteria:

* The HSV serologic status.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any chronic drug therapy to be continued during the study period.
* Receipt of live attenuated vaccines within 30 days of study vaccine administration.
* Receipt of medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) or allergy treatment with antigen injections within 14 days of study vaccine administration.
* Prior receipt of the adjuvant or any of its components being used in this study.
* Previous vaccination against CMV.
* History of recurrent herpes simplex infection (more than 1 episode per year).
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* Hepatitis B infection or hepatitis C infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness including but not limited to diabetes mellitus and thyroid disease
* History of any neurologic disorders or seizures except people with febrile convulsions before the age of 5.
* History of malignancy
* Acute disease at the time of enrollment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Decreased renal function
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of chronic alcohol consumption and/or drug abuse.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02-22 (Actual); Primary Completion 2008-08-27 (Actual); Study Completion 2008-08-27 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general AEs. | During a 7 days follow-up after each vaccination
Occurrence, intensity and relationship to vaccination of unsolicited AEs. | During a 31 days follow-up period after each vaccination
Occurrence and relationship to vaccination of any SAEs. | Throughout the study period
Haematological and biochemical parameters. | At months 0, 1, 2, 6, 7 12 and 24

SECONDARY OUTCOMES:
Anti-gB antibody avidity in all groups; | At months 0, 1, 2, 6, 7 12 and 24
Neutralizing anti-cytomegalovirus (CMV) antibody response in all groups | At months 0, 1, 2, 6, 7, 12 and 24;
Anti-CMV tegument proteins antibody response in all groups; | At months 0, 1, 2, 6, 7, 12 and 24;
Frequencies of CD4/CD8 T-cells with antigen-specific IFN-g, IL-2, TNF-a and/or CD40L secretion/expression to gB as determined by ICS in all groups; | At months 0, 1, 2, 6, 7, 12 and 24
Anti-Herpes simplex virus (HSV) gD antibody response in all groups. | At months 0, 1, 2, 6, 7, 12 and 24
Anti-glycoprotein B (gB) antibody concentrations in all groups; | At months 0, 1, 2, 6, 7, 12 and 24;
Anti-CMV Western Blot in all groups. | At months 0, 1, 2, 6, 7, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Wilrijk

REFERENCES:
- See also: Results for study 108890 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/108890?search=study&b%22b''%22#rs